CLINICAL TRIAL: NCT06745713
Title: The Effectiveness of E-Learning Application Developed For Chest Tube Care in Nursing Students
Acronym: E-GTBYEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Collaborators: Gazi University Scientific Research Unit (Unknown); Atılım University (Other)
Responsible Party: Principal Investigator, Sevil Güler, Prof. Dr., Gazi University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Other
Other Study IDs: E-770082166-302.08.01-509027
Record Dates: First submitted 2024-12-03; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: E-learning; Nursing Care; Chest Tube; Nursing Education
Keywords: chest tube care; e-learning; nursing care; nursing students; clinical reasoning

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: In order to blind the students, the information about which group they were in was not shared with the students, and the students were informed that training on chest tube care management would be given and tests would be applied through the e-learning application. In addition, the students were informed that the contents of the 'Chest Tube Care Management Training Programme' would be opened to everyone at different times, and that the time of opening the tests and training content was determined by the e-learning application itself. The training content was opened to the control group after the post-test data were collected. Thus, blinding of the participant students was ensured. The researcher who recorded all the data obtained as a result of the study in the statistics programme and the person who made the statistical analyses of the data did not know which groups were the experimental or control groups. While analysing the statistical data, the statistician and the researcher knew.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): They completed the chest tube care management training programme which includes 5 modules, 4 case scenarios and interactive questions on www.gtbyep.com website.
  Interventions: Other: Turkish- Computer System Usability Questionnaire Short Version; Other: Student Information Form; Other: Clinical Reasoning Readiness Scale for Nursing Students; Other: Self-directed Learning Scale; Other: Chest Tube Care Management Knowledge Test
- Control Group (Active Comparator): The subject content of chest tube care management in the nursing education curriculum was given. After the pre- and post-tests were completed in the training programme in which the experimental group was included, the control group was also included in the training programme on www.gtbyep.com. The control group also completed the training content as applied to the experimental group.
  Interventions: Other: Student Information Form; Other: Clinical Reasoning Readiness Scale for Nursing Students; Other: Self-directed Learning Scale; Other: Chest Tube Care Management Knowledge Test

INTERVENTIONS:
Other: Turkish- Computer System Usability Questionnaire Short Version — Developed in 1995 by Lewis at IBM, the Computer System Usability Questionnaire (CSUQ) is one of the widely used questionnaires in the field of usability. The scale, which was adapted into Turkish by Erdinç in 2013, consists of 13 items in total. It has 4 sub-dimensions: system usefulness (items 1-6), information quality (items 7-9), interface quality (items 10-12) and general satisfaction (item 13). Each item is scored as 1 (Strongly agree) - 7 (Strongly disagree). The Cronbach α of the scale is > .70 and the Cronbach α value for each sub-dimension varies between .73 and .92. A minimum score of 13 and a maximum score of 91 can be obtained from the scale. A low score is defined as good usability, and the higher the score, the lower the usability quality of the system (Erdinç & Lewis, 2013).
  Arms: Experimental Group
Other: Student Information Form — In the form developed by the researchers in line with the literature, a total of 12 questions were included to determine the socio-demographic characteristics of the students (such as age, gender, academic average, whether they provide care to patients with chest tubes, whether they receive training on chest tube care). All participants in the experimental and control groups were applied once as a pre-test.
Other: Clinical Reasoning Readiness Scale for Nursing Students — It is a comprehensive assessment tool developed by Huang Huiman (2018) to determine the clinical reasoning readiness levels of nursing students in Taiwan (Ho et al., 2021; H.-M. Huang et al., 2018). 'Clinical Reasoning Readiness Scale for Nursing Students' consists of 4 sub-dimensions. These sub-dimensions are 'awareness of clinical clues' (4 items), 'verification of clinical problems' (4 items), 'action determination and implementation' (4 items) and 'evaluation and reflection' (4 items). Each sub-dimension contains four items to assess students' clinical reasoning readiness levels. The lowest score that can be obtained from the scale is 16 and the highest score is 80. Responses to the scale are evaluated on a 5-point Likert scale (5=strongly agree, 4=agree, 3=decided, 2=disagree, 1=strongly disagree). Cronbach's α ranged from 0.894 for the total and 0.78 to 0.89 for each sub-dimension. The corrected item-total correlation is between 0.627-0.728. Higher scores indicate higher levels
Other: Self-directed Learning Scale — The original Self-Managed Learning Scale was used as a self-report scale by Lounsbury et. al. (2009). The Turkish adaptation and validity and reliability study of the scale, which shows the extent to which individuals learn autonomously with a one-dimensional structure, was conducted by Demircioğlu, Öge, Fuçular, Çevik, Nazlıgül, and Özçelik in 2018. The scale is 5-point Likert-type and consists of 10 items. For each item, participants are expected to respond according to 1 (Strongly disagree), 2 (Disagree), 3 (No opinion), 4 (Agree) and 5 (Strongly agree). Cronbach's alpha coefficient of the scale is 0.85. In line with the scores obtained from the scale, above average self-directed learning skill means high and below average self-directed learning skill means low (Demircioğlu et al., 2018). Both groups were applied as pre-test and post-test.
Other: Chest Tube Care Management Knowledge Test — It was created by the researchers in line with the evidence in the literature (Abuejheisheh et al., 2021; Basler, 2020; Bertrandt et al., 2019; Charnock & Evans, 2001; El-Senousy, Mahrous, Abd-Al Salam, & Zedan, 2020; Ho et al., 2021; Tarhan et al., 2016; Zisis et al., 2015). The 'Chest Tube Care Management Knowledge Test' was initially prepared as a total of 43 multiple-choice questions, including the headings and subheadings in each session (Abuejheisheh et al., 2021; Malone, 2015). Expert opinions were obtained from 5 faculty members with clinical experience and studies on chest tube care. The experts gave suitability scores to the knowledge test questions one by one on a 4-point Likert-type scale (1: The item is not suitable, 2: The item should be seriously revised, 3: Suitable should be slightly revised, 4: Suitable). In line with the suggestions from the experts, the questions were reorganised and 9 questions were removed. For the remaining 34 multiple-choice questions in the kno

SUMMARY:
This study was conducted to determine the effectiveness of the e-learning application developed for chest tube care in nursing students. Within the scope of this study, the e-learning application developed for chest tube care in nursing students and the effectiveness of this e-learning application were evaluated.

DETAILED DESCRIPTION:
At the beginning of the study, 'Student Information Form', 'Clinical Reasoning Readiness Scale for Nursing Students', 'Self-Managed Learning Scale' and 'Chest Tube Care Management Knowledge Test' were applied to the participants. Then, the students were divided into two groups, 54 in the experimental group and 54 in the control group, and they were provided to enter the 'Chest Tube Care Management E-Learning Application'. The students in the groups were then asked to complete the module containing activities such as videos, short tests, puzzles in the content of the e-learning application opened to them at different times. When the students in the groups completed the module, 'Clinical Reasoning Readiness Scale for Nursing Students', 'Self-Managed Learning Scale' and 'Chest Tube Care Management Knowledge Test' were applied. Participation in this study was voluntary and participants could leave the study at any stage of the study if they wished. The confidentiality of the participant's data was protected and used only for this study.

Hypothesis 1:

H0: There is no significant difference between the chest tube care management knowledge scores of the students using the chest tube care management e-learning application and the control group students.

H1: There is a significant difference between the chest tube care management knowledge scores of the students using the chest tube care management e-learning application and the control group students.

Hypothesis 2:

H0: There is no significant difference between chest tube care management clinical reasoning readiness scale scores of students using chest tube care management e-learning application and control group students.

H1: There is a significant difference between the clinical reasoning readiness scale scores of the students using the chest tube care management e-learning application and the control group students.

Hypothesis 3:

H0: There is no significant difference between the chest tube care management self-directed learning skill levels of the students using the chest tube care management e-learning application and the control group students.

H1: There is a significant difference between the chest tube care management self-directed learning skill levels of the students using the chest tube care management e-learning application and the control group students.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* To be able to understand and speak Turkish,
* To be enrolled in the 3rd year of the Nursing Department,
* Taking Surgical Diseases Nursing course for the first time,
* To be able to access Internet,
* Voluntary acceptance to participate in the research.

Exclusion Criteria:

* Notifying that he/she wants to leave the research at any stage of the research,
* They did not participate in any of the steps of the e-learning application such as pre-test, watching the videos, post-test, evaluation activities, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
Clinical Reasoning Readiness Scale for Nursing Students | In order to determine the clinical reasoning readiness levels of nursing students, it was applied to the students in the experimental and control groups before the application started and immediately after the application was completed.
  It is a comprehensive assessment tool developed by Huang Huiman (2018) to determine the clinical reasoning readiness levels of nursing students in Taiwan (Huang et al., 2023). 'Clinical Reasoning Readiness Scale for Nursing Students' consists of 4 sub-dimensions. These sub-dimensions are 'awareness of clinical clues' (4 items), 'verification of clinical problems' (4 items), 'action determination and implementation' (4 items) and 'evaluation and reflection' (4 items). Each sub-dimension contains four items to assess students' clinical reasoning readiness levels. The lowest score that can be obtained from the scale is 16 and the highest score is 80. The responses to the scale are evaluated on a 5-point Likert scale (5=Strongly agree, 4=Agree, 3=Unsure, 2=Disagree, 1=Strongly disagree). Cronbach's α ranged from 0.894 for the total and 0.78 to 0.89 for each sub-dimension. The corrected item-total correlation is between 0.627-0.728.
Self-directed Learning Scale | The Self-Managed Learning Scale was administered to the students in the experimental and control groups before and immediately after the implementation of the study.
  The original Self-Managed Learning Scale was used by Lounsbury et al. (2009) as a self-report scale. The Turkish adaptation and validity and reliability study of the scale, which assesses the extent to which individuals learn autonomously with a one-dimensional structure, was conducted by Demircioğlu, Öge, Fuçular, Çevik, Nazlıgül, and Özçelik in 2018. The scale is 5-point Likert-type and consists of 10 items. For each item, participants are expected to respond according to 1 (Strongly disagree), 2 (Disagree), 3 (No opinion), 4 (Agree) and 5 (Strongly agree). Cronbach's alpha coefficient of the scale is 0.85. In line with the scores obtained from the scale, above average self-managed learning skill means high and below average self-managed learning skill means low (Demircioğlu et al., 2018). In this study, the cronbach alpha coefficient of 'Self-Managed Learning Scale' was found to be 0.915 in the pre-test and 0.890 in the post-test.
Chest Tube Care Management Knowledge Test | The Chest Tube Care Management Knowledge Test was administered to the students in the experimental and control groups before and immediately after the implementation of the study.
  The researchers created it in line with the evidence in the literature, including questions on Chest Tube Care Management (Abuejheisheh et al., 2021; Basler, 2020; Bertrandt et al., 2019). The 'Chest Tube Care Management Knowledge Test' was initially prepared as a total of 43 multiple-choice questions including the headings and subheadings in each session (Abuejheisheh et al., 2021; Malone, 2015). Expert opinions were obtained from 5 faculty members with clinical experience and studies on chest tube care. The experts gave suitability scores to the knowledge test questions one by one on a 4-point Likert-type scale (1: The item is not suitable, 2: The item should be seriously revised, 3: Suitable should be slightly revised, 4: Suitable). In line with the suggestions from the experts, the questions were reorganized and 9 questions were removed.

SECONDARY OUTCOMES:
Turkish- Computer System Usability Questionnaire short version | It was applied to the students in the experimental group of the research after the implementation of the research was completed.
  Developed in 1995 by Lewis at IBM, the Computer System Usability Questionnaire (CSUQ) is one of the widely used questionnaires in the field of usability. The scale, which was adapted into Turkish by Erdinç in 2013, consists of 13 items in total. It has 4 sub-dimensions: system usefulness (items 1-6), information quality (items 7-9), interface quality (items 10-12) and general satisfaction (item 13). Each item is scored as 1 (Strongly agree) - 7 (Strongly disagree). The Cronbach α of the scale is > .70 and the Cronbach α value for each sub-dimension varies between .73 and .92. A minimum score of 13 and a maximum score of 91 can be obtained from the scale. A low score is defined as good usability, and the higher the score, the lower the usability quality of the system (Erdinç & Lewis, 2013). In this study, Cronbach's alpha value of the scale was found to be 0.981.
Chest Tube Care Management Training Programme Evaluation Form | It was applied to the students in the experimental group of the research after the implementation of the research was completed.
  This form was created by the researcher in line with the literature (Pires, 2023; Yüksel & Kösterelioğlu, 2023). In order to evaluate the Chest Tube Care Management Training Programme, it was evaluated by SWOT (Strengths, Weaknesses, Opportunities and Threats) analysis. In this direction, the researchers created 23 suggestions for the strengths of the training programme, 6 suggestions for the weaknesses, 8 suggestions for opportunities and 3 suggestions for threats. The form includes a total of 40 propositions in 11-point Likert type. The students were asked to give a score between 0 and 10 according to their level of agreement with each proposition (0 - I do not agree at all, 1 - I agree very little, 10 - I completely agree). The form also includes an open-ended question about the strengths, weaknesses, opportunities and perceived threats of the training programme under each heading, with the option 'Other'.

OTHER OUTCOMES:
Student Information Form | The Student Information Form was applied to all students in the experimental and control groups who agreed to participate in the study once before the start of the study.
  The form, which was developed by the researchers in line with the literature, included a total of 12 questions to determine the socio-demographic characteristics of the students (such as age, gender, academic average, whether they provide care for patients with chest tubes, whether they receive training on chest tube care).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data supporting this study are not publicly available due to ethical reasons but the datasets used and/or analyzed during the current study are available by emailing sevil.guler@gazi.edu.tr upon reasonable request.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 2 years after the publication of results
Access Criteria: They will be able to access via e-mail to sevil.guler@gazi.edu.tr.